The effects of magnesium sulphate on intraoperative blood loss in meningioma patient undergoing craniotomy with tumor removal: A prospective randomized study.

NCT number: NCT03558516

**Document date: 1 August 2018** 

## Statistical Analysis Plan

The collected data will be analyzed by Statistical Package for the Social Sciences (SPSS) software version 18.0 (SPSS Inc., Chicago, IL, USA). Data will be described in terms of frequencies (number and percent of cases), mean ± standard deviation, median (range) when appropriate. Chi-square or Fisher's exact test will be used for comparing categorical data. Student's t-test will be used for comparing continuous data with normal distribution.

Comparison of nonparametric variables will be done using Mann-Whitney test. The p-value < 0.05 will be considered statistical significance.